CLINICAL TRIAL: NCT04746729
Title: Health Effects of CArdiac FluoRoscopy and MOderN RadIotherapy in PediatriCs - Radiotherapy (HARMONIC-RT)
Brief Title: Health Effects of CArdiac FluoRoscopy and MOderN RadIotherapy in PediatriCs - Radiotherapy
Acronym: HARMONIC-RT
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Barcelona Institute for Global Health (Other); The West German Proton Therapy Centre, Essen (Unknown); Gustave Roussy, Cancer Campus, Grand Paris (Other); Centre Francois Baclesse (Other); KU Leuven (Other); University of Aarhus (Other); Princess Maxima Center for Pediatric Oncology (Other); University Medical Center Groningen (Other); Stockholm University (Other); National Research Council, Institute of Clinical Physiology, Italy (Other); University of Zurich (Other); Commissariat A L'energie Atomique (Other Government); Luxembourg Institute of Science and Technology (Other); University Hospital, Essen (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: C20-01; 2020-A01037-32/1 (Registry Identifier: ID RCB)
Record Dates: First submitted 2020-09-14; First posted 2021-02-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Neoplasms
Keywords: Radiotherapy; Oncology; Paediatrics; Late toxicities; Radiation-induced neoplasms; Radiation-induced vascular damages; Radiation-induced cardiac damages; Radiation-induced endocrine damages; Quality of life; Social outcomes; External beam radiotherapy; Photon therapy; Proton therapy; Cohort; Registry
MeSH Terms: conditions — Neoplasms; Neoplasms, Radiation-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — blood plasma; blood serum; lymphocytes; saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of the HARMONIC-RT study is to evaluate late health and social outcomes of contemporary techniques of external beam radiotherapy in paediatric patients, based on the setting-up of a European, long-term registry complemented by a biobank.

DETAILED DESCRIPTION:
Specific objectives:

* To develop the infrastructure and instruments for setting-up a European, long-term registry of paediatric patients treated with contemporary techniques of modern external radiotherapy;
* To assess the incidence and severity of late health outcomes, primarily endocrine dysfunctions, cardiovascular toxicities, neurovascular damages, and subsequent primary neoplasms, in relation to the dose-volume distribution to non-targeted organs and tissues, radiation delivery technique and beam quality factors, and potential modifying factors (i.e. age at exposure, genetic predispositions, comorbidities, and systemic treatments including chemotherapy, targeted therapy, immunotherapy and hormonal drugs) that may underlie differences in individual susceptibility for these outcomes ;
* To assess societal aspects of advances in radiotherapy, primarily health-related quality of life and academic achievement, in paediatric patients treated with modern external radiotherapy techniques.

Secondary scientific objectives:

* To assess multidimensional fatigue in paediatric patients treated with modern external radiotherapy techniques, and identify clinical and therapeutic determinants of fatigue;
* To improve estimation of patient-specific doses to the whole body and non-targeted organs and substructures from different radiotherapy delivery techniques;
* To investigate radiation-induced cellular responses and biological mechanisms related to the occurrence of vascular diseases and subsequent primary neoplasms in samples of blood and saliva ; to identify biomarkers of susceptibility and health effects ; to evaluate differences in disease biomarkers in relation to the radiation delivery technique and beam quality factors ; to explore the relevance of the use of saliva as a biosampling method for paediatric cohorts regarding feasibility and the quality and reproducibility for different measured biomarkers.

Secondary strategic objectives:

* To promote sustained collaborative research activities for improvement of patient care, and inform health care providers and policy makers on the clinical and social impact of advances in radiotherapy in paediatric settings;
* To serve as a pilot for a future long-term pan-European registry of children and adolescents treated with particle and photon beam therapy, including a biobank of saliva and blood samples collected before and after treatment;
* To contribute in future collaborative projects with existing cohorts or registries in Europe
* To contribute in future international research studies on late outcomes of modern radiotherapy techniques for management of paediatric cancers

Funding: The HARMONIC project has received funding from the Euratom research and training programme 2014-2018 under grant agreement No 847707.

ELIGIBILITY:
Retrospective inclusion of study participants

Inclusion Criteria:

* First external beam radiation therapy (EBRT) started in 2000 or after for management of a first primary neoplasm
* Age under 22 years at the time of first EBRT initiation
* Radiation treatment plan (first EBRT) stored in DICOM format
* Usual residency in the country of EBRT to enable a long-term follow-up

Exclusion Criteria:

* Patients with poor prognosis (e.g. diffuse pontine glioma or high grade glioma) at first EBRT initiation
* Prior external or internal radiation therapy
* Patients who refused to participate in the study

Prospective inclusion of study participants

Inclusion Criteria:

* Scheduled first EBRT for management of a first primary neoplasm
* Age under 22 years at the time of scheduled first EBRT
* Radiation treatment plan stored in DICOM format
* Affiliate or beneficiary of health insurance (or any required equivalent as defined in applicable national law)
* Usual residency in the country of EBRT to enable a long-term follow-up
* Signed informed consent/assent

Exclusion Criteria:

* Patients with poor prognosis (e.g. diffuse pontine glioma or high grade glioma)
* Prior external or internal radiation therapy;
* Protected adults (persons under curatorship, tutorship / individuals under guardianship by court order, persons deprived of their liberty)
* Adult/parent(s)/legal representative(s) who cannot read or understand the informed consent in the applicable language(s) in the country of EBRT

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, adolescents and young adults treated with external beam radiation therapy for a first primary neoplasm
Sampling Method: Non-Probability Sample
Enrollment: 2670 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2040-09-30 (Estimated); Study Completion 2040-09-30 (Estimated)

PRIMARY OUTCOMES:
Endocrinopathies | up to 20 years after RT
  Late health outcomes
Cardiovascular diseases | up to 20 years after RT
  Late health outcomes
  * Neurovascular diseases
  * Second and subsequent primary neaoplasms
Neurovascular diseases | up to 20 years after RT
  Late health outcomes
Second and subsequent primary neaoplasms | up to 20 years after RT
  Late health outcomes
Health-related quality of life (physical, emotional, social, and school functioning) assessed by the PedsQL™ core scale (validated questionnaire) | up to 10 years after radiation therapy or attained age 25 years, whichever occurs first
  Late social outcomes
Academic achievement | up to 10 years after radiation therapy or attained age 25 years, whichever occurs first
  Late social outcomes

SECONDARY OUTCOMES:
Dysfunctions in endocrine hormone levels | up to 10 years after radiation therapy
  measured as:
  1. insulin-like growth factor-1,
  2. anterior pituitary hormones (GH, ACTH, TSH, LH, FSH),
  3. thyroid hormones (fT3, fT4),
  4. sexual hormones
Changes in blood markers of cardiovascular diseases | up to 10 years after radiation therapy
  measured as blood markers (incl. troponin, BNP, CPK)
Changes in imaging markers of cardiovascular diseases | up to 10 years after radiation therapy
  measured as cardiac echography parameters (incl. ejection fraction, diastolic function)
Changes in imaging markers of neurovascular damages | up to 5 years after radiation therapy
  measured as scoring of large and small vessel damages
Changes in blood/saliva markers of protein activation relating to vascular damages | up to 1 year after radiation therapy
  measured as signal quality of protein activity
Changes in blood/saliva markers of oxidative stress response | up to 1 year after radiation therapy
  measured as markers of oxidative stress (incl. 8-oxo-dG, SOD2, DNA repair enzymes)
Changes in blood/saliva markers of inflammatory response | up to 1 year after radiation therapy
  Inflammatory markers (incl. PTX3, CRP, NF-kB, IL-1 and IL10)
Changes in blood/saliva markers of carcinogenesis | up to 1 year after radiation therapy
  Markers of carcinogenesis (incl. leukocyte telomere length, mitochondrial DNA copy number, circulating microRNA)
Multidimensional fatigue (general, sleep/rest, and cognitive fatigue) | up to 10 years after radiation therapy or attained age 25 years, whichever occurs first
  PedsQL™ multidimensional fatigue scale (validated questionnaire)
Clinical events other than those mentioned as primary outcomes | up to 20 years after radiation therapy
  Late morbidity
All-cause and cause-specific mortality | up to 20 years after radiation therapy
  Late mortality

CONTACTS AND LOCATIONS:
Overall Officials: Beate Timmermann, MD, Principal Investigator — UK Essen; Neige Journy, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Stéphanie Bolle, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Isabelle Thierry-chef, PhD, Study Chair — Barcelona Institute for Global Health
Locations (5):
- KU Leuven, Leuven, Belgium
- Aarhus University hospital, Aarhus, Denmark
- France (2):
  - Centre Régional François Baclesse, Caen
  - Gustave Roussy, Villejuif
- University Hospital Essen, The West German Proton Therapy Centre Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Journy N, Bolle S, Brualla L, Dumas A, Fresneau B, Haddy N, Haghdoost S, Haustermans K, Jackson A, Karabegovic S, Lassen-Ramshad Y, Thariat J, Wette MR, Botzenhardt S, De Wit I, Demoor-Goldschmidt C, Christiaens M, Hoyer M, Isebaert S, Jacobs S, Henriksen LT, Maduro JH, Ronckers C, Steinmeier T, Uyttebroeck A, Van Beek K, Walsh L, Thierry-Chef I, Timmermann B. Assessing late outcomes of advances in radiotherapy for paediatric cancers: Study protocol of the "HARMONIC-RT" European registry (NCT 04746729). Radiother Oncol. 2024 Jan;190:109972. doi: 10.1016/j.radonc.2023.109972. Epub 2023 Nov 2. No abstract available. PMID 37922994
- See also: Project's website — https://harmonicproject.eu/